CLINICAL TRIAL: NCT02674165
Title: Evaluation of Haitian American Responsible Teens
Acronym: HART
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Nicole Prudent, Associate Clinical Professosr of Pediatrics, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H30298
Record Dates: First submitted 2016-01-27; First posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Sexual Behavior
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The pregnancy prevention intervention to be tested is an adaptation of Becoming a Responsible Teen (BART), an evidence-based (proven to work by research) HIV prevention curriculum designed primarily for African American adolescents, ages 14-18, in community-based settings.
  The culturally-adapted version HART consists of nine sessions, lasting about 2 hours each, and includes interactive group discussions and role plays that are -performed by adolescents. Unlike BART, one PTSD awareness session has been added to address what happens to people who have been exposed to mental trauma and natural disasters.
  Interventions: Behavioral: HART
- Control or nutrition (No Intervention): Nutrition/fitness curriculum will teach students about ingredients in food that are good for the body and will keep it in good health

INTERVENTIONS:
Behavioral: HART — Skills based sexual education intervention plus PTSD awareness
  Arms: Intervention

SUMMARY:
The Haitian American Responsible Teen (HART) afterschool program, a cultural adaptation of the BART curriculum, will provide an HIV/AIDS curriculum adapted to Haitian students that consists of eight sessions lasting approximately two hours each over a twelve- week period. The comparison group will receive a nutrition intervention during the same time period. The primary goals of the evaluation are to determine the effectiveness of the HART program on delaying initiation of sexual intercourse, reducing number of sexual partners, and increasing "abstinent" behavior and contraception use among those who were sexually experienced at baseline.

Over a five semester period, the programs will be implemented in 7 or more schools in the greater Boston area, with offerings in the fall, the spring and summer, among approximately 780 male and female Haitian students. The programs will recruit 9th & 10th grade Haitian students who will range in age from 13 to 19 years old. We will implement a randomized controlled trial in which each semester, students within schools will be stratified by gender and then randomly assigned to participate in the HART or the nutrition condition. Students will be recruited annually and enrolled until the summer of 2015. During the spring and summer of 2012, 120 youth will be randomly assigned to a treatment condition. During year three, 180 youth will be randomly assigned to condition each semester (360 youth total during Year 3). During year four, 180 youth will be randomly assigned in the first semester, and 120 youth will be randomly assigned in the second semester (300 youth total during Year 4). The number of times student-level randomization will occur and the number of groups formed will vary depending on the size of the 9th and 10th grade Haitian population served in each school.

DETAILED DESCRIPTION:
This is an intervention with an evaluation component. In each school, students will have equal chance to participate in the sex education class or in the nutrition education class. Each participating school will have two (2) groups:

* The intervention group which will receive the HART sex education curriculum.
* The comparison group which will receive a nutrition education curriculum. There will be one PTSD awareness session for both groups.. This session will be provided by mental health professionals from the Haitian Mental Health Network. Each group will consist of about 13-15 student participants, with the groups meeting each week on specific week days. In addition to the ten-week curriculum, there will be sessions at the beginning and end of the cycle to administer the pre- and post-test questionnaires. The 12-week cycle will be repeated 2-3 times through the school year.

ELIGIBILITY:
Inclusion criteria

1. Haitian descent
2. 13 to 19 years of age
3. 9th and 10th grade
4. Having signed assent and parental consent forms
5. Willingness to participate in the pretest survey

Exclusion criteria

1. Not of Haitian descent
2. Age greater than 19 years
3. Under 13 years of age
4. Cognitive impairment
5. Not having signed assent and parental consent forms
6. Not willingness to participate in the pretest survey

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 637 (Actual)
Dates: Start 2012-04; Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
HIV knowledge measured by having a statistically significant difference between treatment and control participants, in proportion of true or false statements about HIV transmission, prevention and cure that are accurately identified. | One week after the intervention ended
  This outcome is collected at one week post intervention using a quantitative self-administered survey. Pre-test measures and key demographic data e.g. age, gender and other covariates of prognostic significance that are found not to have a balanced distribution between the treatment and control are adjusted for using multivariate analysis to increase precision of treatment effect measure

SECONDARY OUTCOMES:
Three- cognitive constructs that are causally related with HIV knowledge within the "Information Motivation and Behavioral Skills" framework.. Our study includes : 3 measures of Personal motivation | One week after the intervention ended
  1. A statistically significant posttest difference between treatment and control in proportion of participants reporting definite intent to have sex next year
  2. A statistically significant posttest difference between treatment and control in proportion of participants reporting a definite intent to use condom if have sex in next year
  3. A statistically significant posttest difference between treatment and control in proportion of participants reporting definite intent to use birth control if have sex in next year
4 measures of Social motivation for preventive behavior | One week after the intervention ended
  A statistically significant posttest difference between the treatment and control in proportion of participants reporting not being embarrassed to buy, use, talk about condoms b) A statistically significant posttest difference between the treatment and control in Proportion of participant reporting condom effectiveness to prevent HIV c) A statistically significant posttest difference between the treatment and control in proportion reporting condom effectiveness to prevent pregnancy d) A statistically significant posttest difference between the treatment and control in proportion of participants reporting not believing that condom purchase is a regulation for youth under the age of 16.
4 measures of Behavioral skills of avoiding risky social situations that could engage in risky sexual behavior. | One week after the intervention ended
  1. A statistically significant posttest difference between the treatment and control in Proportion of participants reporting being alone 3 or more times in the last 3 months with someone very attracted to
  2. A statistically significant posttest difference between the treatment and control in proportion of participants reporting being alone 3 or more times in the last 3 months kissing and touching someone really liked
  3. A statistically significant posttest difference between the treatment and control in proportion of participant reporting being alone 3 or more times in the last 3 months with someone really liked and laid down on a couch or bed
  4. A statistically significant posttest difference between the treatment and control in proportion of participants reporting being alone 3 or more times in the last 3 months, at a party where there were no adults in the house

IPD SHARING:
Plan to Share IPD: No